CLINICAL TRIAL: NCT04327661
Title: Motion Syros: A Randomized, Double-blind, Placebo-controlled Study to Investigate the Efficacy of Tradipitant in Subjects Affected by Motion Sickness During Travel
Brief Title: Motion Syros: A Study to Investigate the Efficacy of Tradipitant in Subjects Affected by Motion Sickness
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VP-VLY-686-3401
Record Dates: First submitted 2020-03-26; First posted 2020-03-31 (Actual); Results first posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-11

CONDITIONS: Motion Sickness
MeSH Terms: conditions — Motion Sickness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Tradipitant High Dose (Experimental)
  Interventions: Drug: Tradipitant
- Tradipitant Low Dose (Experimental)
  Interventions: Drug: Tradipitant
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tradipitant — Oral Capsule
  Arms: Tradipitant High Dose; Tradipitant Low Dose
Drug: Placebo — Oral Capsule
  Arms: Placebo

SUMMARY:
A multi-center, randomized, double-blind, placebo-controlled study to investigate the efficacy of tradipitant in subjects affected by motion sickness during travel

ELIGIBILITY:
Inclusion Criteria:

* History of motion sickness
* Age 18-75

Exclusion Criteria:

* Nausea-inducing disorder other than motion sickness
* BMI>40
* History of intolerance and/or hypersensitivity to Neurokinin-1 Receptor antagonists

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Pacific Research Network, LLC, San Diego, California
  - Santa Monica Clinical Trials, Santa Monica, California
  - Gulfcoast Psychiatric Associates, Fort Myers, Florida
  - Harmony Clinical Research, North Miami Beach, Florida
  - Avita Clinical Research, Tampa, Florida
  - Beacon Clinical Research, Quincy, Massachusetts
  - Manhattan Medical Research, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Polymeropoulos VM, Kiely L, Bushman ML, Sutherland EB, Goldberg AR, Pham AX, Miller CR, Mourad R, Davis TR, Pham NV, Morgan DB, Giles AK, Xiao C, Polymeropoulos CM, Birznieks G, Polymeropoulos MH. Motion Syros: tradipitant effective in the treatment of motion sickness; a multicenter, randomized, double-blind, placebo-controlled study. Front Neurol. 2025 Mar 4;16:1550670. doi: 10.3389/fneur.2025.1550670. eCollection 2025. PMID 40103934

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tradipitant High Dose | Tradipitant Low Dose | Placebo
Started | 121 | 123 | 122
Completed | 120 | 123 | 122
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tradipitant High Dose | Tradipitant Low Dose | Placebo | Total
Number analyzed (Participants) | 121 | 123 | 122 | 366
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (14.84) | 49.6 (14.40) | 48.6 (13.48) | 48.6 (14.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 82 | 75 | 244
  Male | 34 | 41 | 47 | 122
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 12 | 14 | 40
  Not Hispanic or Latino | 99 | 102 | 105 | 306
  Unknown or Not Reported | 8 | 9 | 3 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 2 | 3
  Asian | 7 | 9 | 11 | 27
  Black or African American | 10 | 5 | 5 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  White | 103 | 105 | 102 | 310
  Other | 0 | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 121 | 123 | 122 | 366
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: Population does not include withdrawn subjects
  kg/m^2
    number analyzed (Participants) | 120 | 123 | 122 | 365
    (all) | 26.785 (4.6327) | 27.299 (4.9265) | 28.037 (5.1835) | 27.377 (4.9342)

OUTCOME MEASURES:

1. Primary Outcome: Prevention of Vomiting Measured by Vomiting Assessment (VA)
Description: Prevention of vomiting measured by Vomiting Assessment (VA) score in tradipitant high dose. The VA is a 1-item questionnaire to objectively measure the incidence of emesis. Participants will indicate whether or not they have vomited. The Count of Participants indicates participants who vomited.
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Groups:
- Tradipitant High Dose; Tradipitant Low Dose; Placebo: Oral Capsule
Arm/Group | Tradipitant High Dose | Tradipitant Low Dose | Placebo
Number analyzed (Participants) | 120 | 123 | 122
Participants | 22 | 24 | 54

ADVERSE EVENTS:
Time Frame: Adverse Events were recorded from time of randomization until the end of study visit, up to 7 days.
Arm/Group | Tradipitant High Dose | Tradipitant Low Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/120 | 0/123 | 0/122
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/123 | 0/122
Other Adverse Events (participants affected / at risk) | 26/120 | 20/123 | 4/122
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tradipitant High Dose (N=120) | Tradipitant Low Dose (N=123) | Placebo (N=122)
Headache (Nervous system disorders) | 10 | 7 | 3
Somnolence (Nervous system disorders) | 10 | 8 | 1
Fatigue (General disorders) | 10 | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-07): https://cdn.clinicaltrials.gov/large-docs/61/NCT04327661/Prot_SAP_000.pdf